CLINICAL TRIAL: NCT02069496
Title: Drug Use Investigation for Arepanrix® (H1N1)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114128
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2012-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — arepanrix

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects who receive Arepanrix®: Subjects who receive Arepanrix® as per routine practice
  Interventions: Biological: Arepanrix®

INTERVENTIONS:
Biological: Arepanrix® — Injected according to the prescribing information in the locally approved label by the authorities.

SUMMARY:
This post-marketing surveillance study is designed to collect safety information such as post-vaccination adverse events and adverse reactions from recipients of Arepanrix® (H1N1) Intramuscular Injection.

The following items will be investigated as priority investigation items. <Priority investigation items>

1. Allergic reactions
2. Anaphylaxis

ELIGIBILITY:
Inclusion Criteria:

* Subjects who receive Arepanrix® intramuscular injection for the first time

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects who receive Arepanrix® intramuscular injection for the first time
Sampling Method: Probability Sample
Enrollment: 3405 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The number of recipients who have adverse reactions after injection | 29 days
The number of recipients who have post-vaccination adverse events after injection | 29 days
The number of recipients who have allergic reactions after injection | 29 days
The number of recipients who have anaphylaxis after injection | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Suminobu Ito et al. (2013) Post-marketing Surveillance of AS03-adjuvanted Influenza (H1N1) Vaccine in Japan. Pharma Medica. 31(4):135-141.